CLINICAL TRIAL: NCT04370574
Title: Discovery of Soluble Biomarkers for Pancreatic Cancer Using Innovative All-Patient Inclusive Methodology (PanEXPEL2)
Brief Title: Discovery of Soluble Biomarkers for Pancreatic Cancer Using Innovative All-Patient Inclusive Methodology
Acronym: PanEXPEL2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0191
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Neoplasms
Keywords: Biopsy; Fine-Needle; diagnostic imaging; Endosonography
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Soluble Biomarkers dosage — 1. CytoLyt® fluid will be first processed for routine PDAC diagnosis. In essence, the samples are filtered, tissue fragments and cells are kept for analysis while flow-through is kept until the diagnosis is confirmed. Once this is completed, the samples will be transferred to the lab where the proteins found in the CytoLytR fluid will be precipitated and then solubilized. The protein extracts are stored at -80°C pending proteomic analysis. The remaining CytoLytR fluid supernatant is also stored at - 80°C to be used for metabolomics.
  2. Blood sample will be collected from each patient that underwent diagnostic biopsy. Dry tube for serum analysis will be collected at the time of inclusion during the routine blood test. The serum samples are intended for the validation phase (WP4) and will be exclusively dedicated to this study.

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) remains among cancers with a very poor prognosis (1-year survival <20%). Endoscopic ultrasound with fine needle aspiration (EUS/FNA) is the common examination for all patients with suspicious pancreatic mass. A method was recently developed : it preserves the sanitary sample, named EXPEL, which allows standard pathology examination and OMICS analyzes from the "rinse" liquid. After EUS/FNA in clinical practice, the content of the needle is rinsed in CytoLyt® preservative solution. After cytofiltration, this liquid is systematically discarded.

Based on the EXPEL concept, we hypothesise that this all-patients inclusive approach ("Modified EXPEL" procedure) combined with the methodology to access proteomic and metabolomics information in these original samples will allow us to identify a series of clinically useful marker signatures that will ultimately be measurable, non-invasively, in the patient blood.

DETAILED DESCRIPTION:
Clinical and pathological data will be prospectively collected to obtain 2 subgroups: PDAC and non-PDAC according to the final biopsy diagnosis. A combined quantitative analysis of the proteins and their peptides contained in CytoLyt® will be performed. ROC curves, AUC, sensitivity, specificity, positive predictive value and negative predictive value associated to biomarkers will be calculated to isolate combinations of diagnostic biomarkers. Candidate biomarkers will be validated by immunohistochemistry and multiple reaction monitoring. Prognostic biomarkers will be evaluated by generating 1-year overall survival curves and Cox regression.

The present research, modeled on current practice, employs novel and holistic approach - PANEXPEL methodology - to establish a new repertoire of biomarkers for pancreatic cancer. We intent to provide a comprehensive proteomic and metabolomics biomarker signature that will be measurable in the patient blood using common clinical methods. The potential for translation "from benchside to bedside" is especially high due to the involvement of clinical teams. We expect to propose a combined, robust protein/metabolite biomarker signature that can be rapidly tested in the clinics.

Necessary biological resources: Biological resources will include Cytolyt® and Blood Samples, accompanied by a signed Free and Informed Consent for each included patient.

1. CytoLyt® fluid will be first processed by Pathology Dept. of the CHU for routine PDAC diagnosis. In essence, the samples are filtered, tissue fragments and cells are kept for analysis while flow-through is kept until the diagnosis is confirmed. Once this is completed, the samples will be transferred to the lab where the proteins found in the CytoLytR fluid will be precipitated and then solubilized. The protein extracts are stored at -80°C pending proteomic analysis. The remaining CytoLytR fluid supernatant is also stored at - 80°C to be used for metabolomics.
2. Blood sample will be collected from each patient that underwent diagnostic biopsy. Dry tube for serum analysis 5 ml will be collected at the time of inclusion during the routine blood test (mandatory assessment pre-operative or pre-chemotherapy). The blood sample is centrifuged at 1500xg for 15 minutes while the resulting sera are aliquoted (500μl/aliquot; 4-5 aliquots per patient) and stored at -80°C. These samples will be stored at Biologic Resources Center (CRB Montpellier) that is labelled NF-S-96900 (AFNOR). The serum samples are intended for the validation phase (WP4) and will be exclusively dedicated to this study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pancreatic mass and suspicion of pancreatic ductal adenocarcinoma requiring endoscopic ultrasound with fine needle biopsy

Exclusion Criteria:

* Vulberable person according to L1121-6 of Public health reglementation in France
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with pancreatic mass and suspicion of pancreatic ductal adenocarcinoma requiring endoscopic ultrasound with fine needle biopsy.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Predictive value of each protein contained in Cytolyt® for the positive diagnosis of pancreatic ductal adenocarcinoma | Baseline
  Predictive value of each protein contained in Cytolyt® for the positive diagnosis of pancreatic ductal adenocarcinoma Correlation with positive diagnosis of pancreatic ductal adenocarcinoma and proteins quantity in Cytolyt® samples using ROC curves (sensibility/specificity: Area Under the Curve > 0.85) and binary logistic regression method with controlling for the effects of the co-variates (such as age, disease cTNM stage, and treatment details).

SECONDARY OUTCOMES:
Disease-free survival | One year
  Disease-free survival (percentage of patients without recurrence) .Biomarkers that are prognostically significant on disease free or overall survival in patients with pancreatic cancer, identified using the survival analysis
Disease-free survival | One year
  Biomarkers that are prognostically significant on disease free or overall survival in patients with pancreatic cancer, identified using the survival analysis.
  Disease-free survival (DFS) (time from diagnosis to time of first radiological evidence of local, regional, or distant relapse, or death due to any cause)
Overall survival | One year
  Biomarkers that are prognostically significant on disease free or overall survival in patients with pancreatic cancer, identified using the survival analysis Overall survival at 1 year (percentage of patients alive)
Identification of prognostically significant biomarkers | One year
  Biomarkers that are prognostically significant on disease free or overall survival in patients with pancreatic cancer, identified using the survival analysis.
  Kaplan Meier analysis, logrank test and Cox's proportional hazards regression model to identify biomarkers that are prognostically significant (Hazard ratio (HR) and its 95% confidence interval (CI)

CONTACTS AND LOCATIONS:
Locations (1):
- Uh Montpellier, Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided